CLINICAL TRIAL: NCT01045538
Title: A Phase I/II Study of Vorinostat (Zolinza®) in Combination With Capecitabine (X) and Cisplatin (P) for 1st Line Treatment of Metastatic or Recurrent Gastric Cancer
Brief Title: Study of Vorinostat Plus Capecitabine (X) and Cisplatin (P) for 1st Line Treatment of Metastatic or Recurrent Gastric Cancer: Zolinza+XP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0903
Record Dates: First submitted 2010-01-06; First posted 2010-01-11 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Gastric Cancer; Histone Deacetylase Inhibitor
Keywords: gastric cancer; histone deacetylase inhibitor; 1st line chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Vorinostat; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat plus XP (Experimental): Vorinostat 200~400mg per day on day1-day14 combined with capecitabine 800-1,000mg/m2/dose, BID on day1-day14, and cisplatin 60-80mg/m2 on day 1
  Interventions: Drug: Vorinostat, capecitabine, and cisplatin

INTERVENTIONS:
Drug: Vorinostat, capecitabine, and cisplatin — Vorinostat 200~400mg per day on day1-day14 combined with capecitabine 800-1,000mg/m2/dose, BID on day1-day14, and cisplatin 60-80mg/m2 on day 1
  Other Names: Zolinza, and xeloda

SUMMARY:
There is scientific rationale for exploring the role of vorinostat, histone deacetylase inhibitor with capecitabine (X) and cisplatin (P), one of standard chemotherapy in patients with advanced gastric cancer. XP is a new standard of care in advanced gastric cancer (AGC) and vorinostat is a novel targeted agent that prevents tumor cell proliferation, survival and angiogenesis through histone deacetylase inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable or metastatic advanced gastric adenocarcinoma
* Completion of adjuvant chemotherapy 6 months before the study, or no previous chemotherapy
* Age 18 to 70 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 2 or less
* Estimated life expectancy of more than 3 months
* Presence of measurable or evaluable disease
* Adequate bone marrow function (ANC >1,500/µL and platelets>100,000/µL),
* Adequate renal function: creatinine < 1 x upper normal limit (UNL) or creatinine clearance 60ml/min or less
* Adequate hepatic function: bilirubin < 1.5 x UNL, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) levels < 2.5 x UNL (< 5 x upper limit of normal for patients with liver involvement of their cancer), alkaline phosphatase < 5 x UNL (except in case of bone metastasis without any liver disease)
* Written informed consent

Exclusion Criteria:

* Prior exposure to any histone deacetylase (HDAC) inhibitor (however, valproic acid would be allowed if a 30-day wash-off period is provided.)
* Previous adjuvant treatment with capecitabine or platinums
* Contraindication to any drug contained in the chemotherapy regimen
* Other tumor type than adenocarcinoma
* Presence or history of central nervous system (CNS) metastasis
* Gastric outlet or bowel obstruction
* Evidence of serious gastrointestinal bleeding
* Peripheral neuropathy > grade 2
* History of significant neurologic or psychiatric disorders
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Active human immunodeficiency virus (HIV) infection
* Viral hepatitis infections
* Other serious illness or medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Phase 1 - maximum tolerated dose, Phase 2 - response rate | 3 weeks for maximum tolerated dose, and 6 months for response rate

SECONDARY OUTCOMES:
Toxicity profile | toxicity for each cycle
Progression-free survival | 1 year
  Time from first administration of study drug to disease progression or any cause of death
Overall survival | 1 year
  Time from first administration of study drug to any cause of death

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Budman DR, Meropol NJ, Reigner B, Creaven PJ, Lichtman SM, Berghorn E, Behr J, Gordon RJ, Osterwalder B, Griffin T. Preliminary studies of a novel oral fluoropyrimidine carbamate: capecitabine. J Clin Oncol. 1998 May;16(5):1795-802. doi: 10.1200/JCO.1998.16.5.1795. PMID 9586893
- [Background] Cassidy J, Dirix L, Bissett D, Reigner B, Griffin T, Allman D, Osterwalder B, Van Oosterom AT. A Phase I study of capecitabine in combination with oral leucovorin in patients with intractable solid tumors. Clin Cancer Res. 1998 Nov;4(11):2755-61. PMID 9829739
- [Background] Glimelius B, Ekstrom K, Hoffman K, Graf W, Sjoden PO, Haglund U, Svensson C, Enander LK, Linne T, Sellstrom H, Heuman R. Randomized comparison between chemotherapy plus best supportive care with best supportive care in advanced gastric cancer. Ann Oncol. 1997 Feb;8(2):163-8. doi: 10.1023/a:1008243606668. PMID 9093725
- [Background] Hansen RM. 5-Fluorouracil by protracted venous infusion: a review of recent clinical studies. Cancer Invest. 1991;9(6):637-42. doi: 10.3109/07357909109039875. PMID 1747791
- [Background] Hong YS, Song SY, Lee SI, Chung HC, Choi SH, Noh SH, Park JN, Han JY, Kang JH, Lee KS, Cho JY. A phase II trial of capecitabine in previously untreated patients with advanced and/or metastatic gastric cancer. Ann Oncol. 2004 Sep;15(9):1344-7. doi: 10.1093/annonc/mdh343. PMID 15319239
- [Background] Kim NK, Park YS, Heo DS, Suh C, Kim SY, Park KC, Kang YK, Shin DB, Kim HT, Kim HJ, et al. A phase III randomized study of 5-fluorouracil and cisplatin versus 5-fluorouracil, doxorubicin, and mitomycin C versus 5-fluorouracil alone in the treatment of advanced gastric cancer. Cancer. 1993 Jun 15;71(12):3813-8. doi: 10.1002/1097-0142(19930615)71:123.0.co;2-5. PMID 8508349
- [Background] Kim TW, Kang YK, Ahn JH, Chang HM, Yook JH, Oh ST, Kim BS, Lee JS. Phase II study of capecitabine plus cisplatin as first-line chemotherapy in advanced gastric cancer. Ann Oncol. 2002 Dec;13(12):1893-8. doi: 10.1093/annonc/mdf323. PMID 12453857
- [Background] Koizumi W, Saigenji K, Ujiie S, Terashima M, Sakata Y, Taguchi T; Clinical Study Group of Capecitabine. A pilot phase II study of capecitabine in advanced or recurrent gastric cancer. Oncology. 2003;64(3):232-6. doi: 10.1159/000069313. PMID 12697963
- [Background] Kurdistani SK. Histone modifications as markers of cancer prognosis: a cellular view. Br J Cancer. 2007 Jul 2;97(1):1-5. doi: 10.1038/sj.bjc.6603844. Epub 2007 Jun 26. PMID 17592497
- [Background] Mann BS, Johnson JR, Cohen MH, Justice R, Pazdur R. FDA approval summary: vorinostat for treatment of advanced primary cutaneous T-cell lymphoma. Oncologist. 2007 Oct;12(10):1247-52. doi: 10.1634/theoncologist.12-10-1247. PMID 17962618
- [Background] Park YS, Jin MY, Kim YJ, Yook JH, Kim BS, Jang SJ. The global histone modification pattern correlates with cancer recurrence and overall survival in gastric adenocarcinoma. Ann Surg Oncol. 2008 Jul;15(7):1968-76. doi: 10.1245/s10434-008-9927-9. Epub 2008 May 10. PMID 18470569
- [Background] Weichert W, Roske A, Gekeler V, Beckers T, Ebert MP, Pross M, Dietel M, Denkert C, Rocken C. Association of patterns of class I histone deacetylase expression with patient prognosis in gastric cancer: a retrospective analysis. Lancet Oncol. 2008 Feb;9(2):139-48. doi: 10.1016/S1470-2045(08)70004-4. PMID 18207460